CLINICAL TRIAL: NCT01874756
Title: The Efficacy and Safety of a Selective Estrogen Receptor Beta Agonist (LY500307) for Negative Symptoms and Cognitive Impairment Associated With Schizophrenia
Acronym: Beta
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding ended
Sponsor: Indiana University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Alan Breier, Psychiatrist, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1303010802
Record Dates: First submitted 2013-05-20; First posted 2013-06-11 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Schizophrenia
Keywords: schizophrenia; Estrogen receptor agonist; cognitive impairment; negative symptoms
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — erteberel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LY500307 150mg (Experimental): LY500307 150mg
  Interventions: Drug: LY500307 150mg
- placebo (Placebo Comparator): placebo 6 pills of inactive drug
  Interventions: Drug: Placebo
- LY500307 75mg (Experimental): LY500307 75mg
  Interventions: Drug: LY500307 75mg
- LY500307 25mg (Experimental): LY500307 25mg
  Interventions: Drug: LY500307 25mg

INTERVENTIONS:
Drug: LY500307 150mg — LY500307 150mg daily dose (6 capsules of 25mg) for 8 weeks
  Arms: LY500307 150mg
Drug: LY500307 75mg — LY500307 75mg daily dose (3 capsules of 25mg and 3 capsules of placebo) for 8 weeks
  Arms: LY500307 75mg
Drug: Placebo — 6 placebo capsules daily for 8 weeks
  Arms: placebo
Drug: LY500307 25mg — LY500307 25mg daily dose (1 capsules of 25mg and 5 capsules of placebo) for 8 weeks
  Arms: LY500307 25mg

SUMMARY:
The primary objectives of this application are to determine if the selective ERβ agonist LY500307, when added to antipsychotic medications, improves negative and/or cognitive symptoms in patients with schizophrenia. The specific hypotheses to be tested are to determine if LY500307 is safe and well tolerated in this population and whether it elicits a sufficient efficacy signal to be advanced for further testing in schizophrenia. A two-stage Phase 1b/Phase 2a adaptive ("drop the inferior dose") experimental design is ongoing that combines three studies (clinical dose optimization, cortical target engagement confirmation and efficacy and safety assessment) into a single clinical trial.

Stage 1 was conducted in year 1 and Stage 2 will be conducted in years 2 and 3. The goal of Stage 1 was to identify and advance the highest dose that did not demonstrate a safety signal and had target selectivity as determined by lack of TT suppression. This criteria was fulfilled at both doses, the larger of the two (75 mg/day dose) was advanced to Stage 2. Furthermore, there was no suggestion of ERα receptor activation (i.e., no pattern of TT decreases or feminization AEs) at either dose (25 mg/day and 75 mg/day). A third arm of 150 mg/day was added to Stage 2 for evaluation. Stage 2 results in the following three arms: placebo, 75 mg/day and 150 mg/day. The goals of Stage 2 are to further assess LY500307 doses for safety and target selectivity, confirm cortical target engagement and assess efficacy.

Primary Aim 1: To determine if LY500307 demonstrates cortical target engagement as assessed by fMRI/N-back in frontal-parietal regions. Secondary measures of target engagement are fMRI episodic memory, Pseudo-Continuous Arterial Spin Labeling, Mismatch Negativity/evoked response potentials, Auditory Steady State Response, Auditory P300 and Quantitative EEG (QEEG).

Primary Aim 2: To determine if LY500307 is superior to placebo for one or more of the primary efficacy endpoints: negative symptoms (Negative Symptom Assessment Scale - 16-item total score), working memory (the composite score for the Letter Number Sequencing and Spatial Span tests) and verbal memory (Hopkins Verbal Learning Test).

Primary Aim 3: To determine if LY500307 reduces total testosterone (TT) plasma concentrations, which is indicative of loss of selectivity for ERβ and engagement of ERα, using the following criteria: Decrease in TT plasma concentrations of 50% from baseline in 50% of subjects per arm treated for two consecutive post-randomization values with LY500307 in Stage 1 and Stage 2 of the trial.

Primary Aim 4: To assess the safety of LY500307 by determining if there are SAEs, AEs "probably related to study drug," QTc prolongation, TT suppression (50% reduction from baseline) and to evaluate for other safety signals.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age at study entry
* Male
* DSM IV-TR diagnosis of schizophrenia as confirmed by Structured Clinical Interview for DSM-IV-TR (SCID)
* Outpatient or inpatient status
* Mild to moderate overall disease severity as defined by a CGI-S score of less than or equal to 4 (moderately ill) at randomization
* Moderate levels of negative symptoms as defined by a PANSS negative symptom sub-score greater than or equal to 11.
* Clinical stability as defined by:

  1. No exacerbation of illness leading to an intensification of treatment in the opinion of the investigator within four weeks prior to randomization, and
  2. No change in antipsychotic medication for at least four weeks prior to randomization

Exclusion Criteria:

* Subjects with current acute, serious, or unstable medical conditions, including, but not limited to: inadequately controlled diabetes, asthma, COPD, severe hypertriglyceridemia, recent cerebrovascular accidents, acute systemic infection or immunologic disease, unstable cardiovascular disorders, malnutrition, or hepatic, renal gastroenterologic, respiratory, endocrinologic, neurologic, hematologic, or infectious diseases
* Known or suspected history of prostate cancer, breast cancer, or other clinically significant neoplastic disease (other than squamous cell or basal cell carcinoma of skin)
* Known or suspected history of deep venous thrombosis, stroke, venous thromboembolism, pulmonary embolism, paresis or paralysis that may be thrombogenic in origin
* Subjects currently receiving testosterone replacement therapy or drugs that influence the hypothalamus-pituitary-gonadal axis.
* Subjects who have clinically significant extrapyramidal signs (EPS) as defined by a score of >20 on the Simpson-Angus Scale (SAS)
* Clinically significant electrocardiogram (ECG) abnormality, including, but not limited to, a corrected QT interval (Bazett's; QTcB) >450 msec. Repeat ECGs may be conducted at the discretion of the principal investigator.
* Subjects with known medical history of Human Immunodeficiency Virus positive (HIV+) status
* Subjects with an active seizure disorder
* Subjects with implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, ventriculoperitoneal shunt, or other contraindication to undergoing an MRI scan
* Known IQ less than 70 based on medical history
* Current DSM IV-TR diagnosis of substance dependence (excluding caffeine and nicotine)
* Subjects who test positive for (1) Hepatitis C virus antibody or (2) Hepatitis B surface antigen (HBsAg) with or without positive Hepatitis B core total antibody
* Subjects with moderate to severe renal impairment as defined by creatinine clearance (CrCl) < 60 ml/min (measured by the Cockcroft-Gault equation) at screening. Repeat evaluation may be conducted at the discretion of the Principal Investigator.
* Subjects with hepatic impairment as defined by liver transaminases or total bilirubin > 3 × upper limit of normal (ULN). Repeat evaluation may be conducted at the discretion of the Principal Investigator.
* Subjects considered a high risk for suicidal acts - active suicidal ideation as determined by clinical interview OR any suicide attempt in 30 days prior to screening
* Subjects who have participated in a clinical trial with any pharmacological treatment intervention for which they received study-related medication in the four weeks prior to randomization OR subjects currently receiving treatment (within 1 dosing interval plus four weeks) with an investigational depot formulation of an antipsychotic medication
* Subjects who demonstrate overtly aggressive behavior or who are deemed to pose a substantial risk of danger in the Investigator's opinion

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Breier, MD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - Indiana University Center for NeuroImaging, Indianapolis, Indiana
  - IU Biostatistics, Indianapolis, Indiana
  - Prevention and Recovery Center for Early Psychosis, Indianapolis, Indiana
  - Larue D Carter Memorial Hospital, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | LY500307 25mg | LY500307 75mg | LY500307 150mg
Started | 29 | 10 | 29 | 27
Completed | 28 | 10 | 27 | 21
Not Completed | 1 | 0 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LY500307 25mg | LY500307 75mg | LY500307 150mg | Total
Number analyzed (Participants) | 29 | 10 | 29 | 25 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 10 | 29 | 25 | 93
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.28 (12.27) | 36.64 (12.58) | 37.15 (13.67) | 37.64 (10.21) | 37.07 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 29 | 10 | 29 | 25 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 17 | 6 | 17 | 12 | 52
  White | 11 | 2 | 12 | 13 | 38
  More than one race | 1 | 2 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 10 | 29 | 25 | 93

OUTCOME MEASURES:

1. Primary Outcome: Negative Symptom Changes - Negative Symptom Assessment Scale - 16-item (NSA-16) Total Score
Description: The Negative Symptom Assessment Scale - 16-item (NSA-16) is used to help clinicians rate behaviors (not psychopathology) commonly associated with negative symptoms of schizophrenia. The scale rates subjects on 16 "anchors," is a semi-structured, clinical interview, and each item is rated from 1 to 6. The total score is the sum of the 16 specific items and ranges from 16 to 96; a higher score indicates greater severity of illness. In addition, there is a global rating that represents the overall assessment of a subject's negative symptoms. The rating should not be an average of any particular behavior, but a gestalt of everything observed in the interview.
Time Frame: Baseline, week 2, week 4, week 6, week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LY500307 150mg | Placebo | LY500307 75mg | LY500307 25mg
Number analyzed (Participants) | 25 | 29 | 29 | 10
score on a scale
  Baseline | 42.52 (11.05) | 45.34 (12.03) | 45.93 (13.99) | 46.10 (12.60)
  Week 2 | 40.96 (12.82) | 46.10 (14.68) | 44.82 (11.62) | 47.20 (14.69)
  Week 4 | 41.35 (12.38) | 48.21 (14.32) | 45.30 (12.16) | 45.80 (13.41)
  Week 6 | 43.43 (15.36) | 46.46 (15.64) | 43.19 (11.18) | 44.10 (15.74)
  Week 8 | 42.90 (14.09) | 47.79 (16.26) | 44.12 (12.72) | 44.50 (13.56)

2. Primary Outcome: Working Memory Composite Score Changes
Description: Working memory (composite score of the Wechsler Memory Scale-III: Spatial Span (WMS) and Letter Number Span (LNS) tests). WMS has 2 sections in which a subject recalls increasingly difficult sequences. The total raw score range for both sections is 0-32. The raw score is then converted to a tscore based on normative ranges by age and sex, ranging from 0-100. For both the raw and tscore a higher score reflects better performance.
  LNS consists of 24 increasingly difficult sequences of letters and numbers that a subject is to recall and repeat back in Numeric-Alpha sequential order. The total raw score range is 0-24. The raw score is then converted to a tscore based on normative ranges by age and sex, ranging from 0-100. For both the raw and tscore a higher score reflects better performance.
  The Working Memory composite score is calculated by summing the WMS and LNS tscores, ranging from 0-200, a higher tscore reflects better performance.
Time Frame: Baseline, week 2, week 4, week 6, week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LY500307 150mg | Placebo | LY500307 75mg | LY500307 25mg
Number analyzed (Participants) | 25 | 29 | 29 | 10
score on a scale
  Baseline | 34.76 (12.03) | 33.21 (11.86) | 34.79 (10.90) | 35.70 (14.88)
  Week 2 | 35.70 (10.68) | 36.41 (12.55) | 36.89 (8.94) | 36.50 (13.09)
  Week 4 | 35.30 (13.08) | 35.93 (12.14) | 37.54 (8.66) | 35.90 (13.49)
  Week 6 | 37.13 (11.43) | 36.00 (10.99) | 38.54 (9.63) | 37.20 (13.37)
  Week 8 | 37.86 (11.24) | 38.04 (13.08) | 37.48 (9.18) | 38.00 (12.27)

3. Primary Outcome: Verbal Learning Composite Score Changes
Description: Verbal learning (composite score of the Hopkins Verbal Learning Test-Revised (HVLT-R)). The HVLT-R has 3 trials in which a subject recalls has many words from a list of 12 as they can. The total number recalled for each trial is summed and the score range is between 0-36. The raw score is then converted to a tscore based on normative ranges by age and sex, ranging from 0-100. For both the raw and tscore a higher score reflects better performance.
  The verbal learning composite score is calculated by using the HVLT-R tscore, a higher tscore reflects better performance.
Time Frame: Baseline, week 2, week 4, week 6, week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LY500307 150mg | Placebo | LY500307 75mg | LY500307 25mg
Number analyzed (Participants) | 25 | 29 | 29 | 10
score on a scale
  Baseline | 33.36 (6.60) | 33.93 (5.98) | 34.50 (7.39) | 32.30 (6.63)
  Week 2 | 34.17 (6.97) | 35.41 (8.73) | 37.11 (8.22) | 34.20 (4.87)
  Week 4 | 33.96 (7.04) | 35.11 (7.43) | 37.42 (8.26) | 34.60 (5.52)
  Week 6 | 33.74 (6.78) | 34.44 (7.84) | 34.62 (7.13) | 33.40 (6.28)
  Week 8 | 34.67 (5.63) | 35.54 (7.57) | 37.12 (7.76) | 37.30 (6.17)

4. Primary Outcome: Number of Subjects With Total Testosterone Reduction
Description: Number of subjects with total testosterone reduction, as defined as a decrease in total testosterone plasma concentrations of 50% from baseline for two consecutive post-randomization values
Time Frame: week 2, week 4, week 8
Measure: Number; unit: participants
Arm/Group | LY500307 150mg | Placebo | LY500307 75mg | LY500307 25mg
Number analyzed (Participants) | 25 | 29 | 29 | 10
participants
  Week 2 | 0 | 0 | 0 | 0
  Week 4 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With QTc Prolongation
Description: Number of subjects with QTc prolongation, as defined as any subject with a change from baseline of 60 msec or greater during the active treatment phases
Time Frame: Week 4, Week 8
Measure: Number; unit: participants
Arm/Group | LY500307 150mg | Placebo | LY500307 75mg | LY500307 25mg
Number analyzed (Participants) | 25 | 29 | 29 | 10
participants
  Week 4 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0

6. Primary Outcome: Cortical Target Engagement
Description: To determine if LY500307 demonstrates cortical target engagement as assessed by changes in the N-back in frontal-parietal regions during the MRI.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: beta coefficient
Arm/Group | LY500307 150mg | Placebo | LY500307 75mg | LY500307 25mg
Number analyzed (Participants) | 25 | 29 | 29 | 10
beta coefficient
  Baseline | 0.15 (0.22) | 0.16 (0.22) | 0.27 (0.21) | 0.21 (0.20)
  Week 8 | 0.26 (0.21) | 0.22 (0.22) | 0.31 (0.26) | 0.30 (0.22)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the 8 week time period that subjects were enrolled in the study.
Arm/Group | Placebo | LY500307 25mg | LY500307 75mg | LY500307 150mg
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/10 | 0/29 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/10 | 0/29 | 1/25
Other Adverse Events (participants affected / at risk) | 4/29 | 1/10 | 3/29 | 7/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=29) | LY500307 25mg (N=10) | LY500307 75mg (N=29) | LY500307 150mg (N=25)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematemesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=29) | LY500307 25mg (N=10) | LY500307 75mg (N=29) | LY500307 150mg (N=25)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Increased Urinary Frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Psychotic Exacerbation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT01874756/Prot_SAP_000.pdf